CLINICAL TRIAL: NCT03269396
Title: A Prospective Nonrandomized Study of Laryngeal Allograft Transplantation Clinical Investigation
Brief Title: Laryngeal Allograft Transplantation
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol revision
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David G. Lott, M.D., Consultant-Department of Otolaryngology Head & Neck Surgery/Audiology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-005642; NCI-2024-05947 (Registry Identifier: CTRP (Clinical Trials Reporting Program))
Record Dates: First submitted 2017-08-07; First posted 2017-08-31 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Larynx Stenosis; Larynx Disease; Laryngectomy; Larynx; Larynx Fracture
Keywords: severe laryngotracheal dysfunction
MeSH Terms: conditions — Laryngostenosis; Laryngeal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Larynx Allograft Transplantation (Experimental): Cadaveric laryngotracheal transplantation
  Interventions: Procedure: Larynx Allograft Transplantation

INTERVENTIONS:
Procedure: Larynx Allograft Transplantation — This study is a prospective clinical trial designed to assess the efficacy and safety of laryngeal transplantation. A total of 10 patients will be enrolled over a five-year timeframe. Study length is 5 years.

SUMMARY:
The purpose of this proposed study is to obtain safety and efficacy data on human laryngeal allograft transplantation in an effort to safely use these procedures as a viable reconstructive option for patients with severe laryngeal or laryngotracheal incompetence.

DETAILED DESCRIPTION:
Patients with severe laryngeal or laryngotracheal incompetence without other reconstructive options will be considered for cadaveric laryngotracheal transplantation. Data will be collected from 10 patients and will include length of hospital stay, short-term complications, long-term complications, hospital readmission, return trips to the operating room (OR), rejection episodes and severity, swallowing function, ability to have tracheotomy tube decannulated, voice parameters, pulmonary function, development of anti-donor antibodies, and quality of life scores.

ELIGIBILITY:
Potential subjects for this study include patients with severe laryngeal dysfunction or a previous laryngectomy. For the purposes of this study, severe laryngeal dysfunction is defined as the loss of normal laryngeal function resulting in significant dysphonia, dysphagia, or dyspnea.

Inclusion Criteria:

* Ages 18 years and older
* Male or Female
* One of the following:

  * Severe laryngeal dysfunction as described above
  * Laryngeal stenosis
  * 5 years or longer s/p definitive management for head and neck cancer
  * Laryngeal cancer requiring total laryngectomy in a patient already on immunosuppression
  * Low-grade chondrosarcoma requiring total laryngectomy
* Ability to obtain informed consent from the patient

Exclusion Criteria:

Poor surgical candidacy secondary to poor physical/mental health as determined by a pre-operative medical evaluation

General medical status

* Pregnancy
* Any systemic disease which would alter life expectancy

  * Active neoplastic disease, not considered yet to be cured (Exceptional cases will be considered in case by case discussion)Less than 5 years s/p definitive management for cancer
  * Cancer within the last 5 years (Exceptional cases will be considered in case by case discussion)
  * Obesity (Body Mass Index >29 - 30)(Exceptional cases will be considered on a case by case basis)
  * Cachexia (BMI<18)(Exceptional cases will be considered on a case by case basis) Significant renal dysfunction (Creatinine clearance < 50 ml/min.)
  * Significant hepatic dysfunction
  * Significant kidney damage
  * Unmanageable infections
  * Unable to participate in preoperative exercise training
  * Unable to be weaned to equal or less than 10 mg/day of steroids
  * Untreatable cardiac disease
  * Active neuromuscular disease
  * History of recurrent aspiration or active, unmanageable Gastro-Esophageal Reflux
  * Patients with active connective tissue diseases (exceptions to be considered in a case by case basis)
  * Patients unable to achieve > 600 feet in a 6 minute walk test (exceptions to be considered in a case by case basis)
  * Patients considered having active immunodeficiency disorders (exceptions to be considered in a case by case basis)
  * Multiple co-morbidities that would make transplantation prohibitively risky
* Psychosocial parameters

  * Severe mental retardation, psychosis, depression or organic brain syndrome
  * Uncontrolled diabetes mellitus. Once HbA1C < 7, reevaluate for candidacy.
  * Active substance use within 6 months
  * Active smoking within 6 months
  * Active alcoholism within 6 months
  * Inability to comply with transplant-related management and medical follow-up
  * Any other circumstances that deem the candidate high risk from a psychosocial perspective

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2033-05 (Estimated)

PRIMARY OUTCOMES:
Survival of the allograft at the one-year visit. | 1 year
  Survival of the allograft as indicated by histological rejection grading.

SECONDARY OUTCOMES:
Swallowing without aspiration at the one-year visit. | 1 year
Voice Evaluation | 1 year
  Standard voice evaluation will include voice recordings, acoustic and aerodynamic measurements as compared to baseline measurements.
Pulmonary function | 1 year
  Pulmonary function values within normal range.
Ability to have tracheotomy tube decannulated | 1 year
  Ability to have tracheotomy tube decannulated after successful capping trials.

CONTACTS AND LOCATIONS:
Overall Officials: David G Lott, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Larynx and trachea transplant — https://www.mayoclinic.org/tests-procedures/larynx-trachea-transplant/about/pac-20532544